CLINICAL TRIAL: NCT00914680
Title: Investigation of Efficacy and Tolerability of Magnetic Seizure Therapy in the Treatment of Depression
Brief Title: Berlin Magnetic Seizure Therapy Depression Trial 01
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Malek Bajbouj, Prof. Dr., Charite University, Berlin, Germany
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BEMAST1
Record Dates: First submitted 2009-06-03; First posted 2009-06-05 (Estimated); Last update posted 2018-07-13 (Actual); Status verified 2018-07

CONDITIONS: Unipolar Depression; Bipolar Depression
MeSH Terms: conditions — Depressive Disorder; Bipolar Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MST (Experimental)
  Interventions: Procedure: magnetic seizure therapy

INTERVENTIONS:
Procedure: magnetic seizure therapy — antidepressant treatment with MST

SUMMARY:
This treatment pilot study will investigate clinical efficacy and adverse effects of magnetic seizure therapy (MST) in patients currently experiencing a unipolar or bipolar depressive episode. The investigators will perform add-on tests to assess clinical and cognitive response to treatment. It is hypothesized that MST will have an antidepressant efficacy with a beneficial neurocognitive adverse effect profile.

ELIGIBILITY:
Inclusion Criteria:

* Patient is diagnosed with a severe major depressive episode
* Patient is in a chronic current MDE and/or has had a history of recurrent MDEs
* Patient has not had an acceptable clinical response due to failure with at least 2 antidepressant treatments during the current episode
* Patient has a score > 20 on the HAMD24
* Patient is stable on current psychotropic medication for at least 4 weeks
* Patient is > 25 and < 80 years

Exclusion Criteria:

* Atypical Depression or psychotic depression (according to DSM IV)
* Other relevant psychiatric axis I or axis II diseases
* Relevant neurological diseases
* Relevant cardiac or pulmonary diseases with enhances anesthesiological risk (ASA Score > 3)
* Patient is currently enrolled in another investigational study not associated with the current study
* Patient has a history of, or evidence of, significant brain malformation or significant head injury

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2009-06; Primary Completion 2012-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Clinical Improvement (HAMD) | before, after treatment

SECONDARY OUTCOMES:
Neurocognitive performance | before/after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry, CC15, CBF, Eschenallee 3, Berlin, Germany

REFERENCES:
- See also: Related Info — http://www.charite-psychiatrie.de